CLINICAL TRIAL: NCT00439803
Title: A Single-Site, Phase 1, Double-Blind, Safety and Immunogenicity Trial of an Alphavirus Replicon Vaccine Expressing Cytomegalovirus Genes (AVX601) in Healthy Volunteers
Brief Title: A Clinical Trial of an Alphavirus Replicon Vaccine for Cytomegalovirus (CMV)
Acronym: CMV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AlphaVax, Inc. (Industry)
Responsible Party: Robert A. Olmsted, Ph.D., AlphaVax, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AVX601-001
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Last update posted 2008-11-10 (Estimated); Status verified 2008-11

CONDITIONS: Cytomegalovirus Infections
Keywords: CMV; cytomegalovirus; Alphavirus
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- T1 (Active Comparator)
  Interventions: Biological: AVX601
- C1 (Placebo Comparator)
  Interventions: Biological: Placebo
- T2 (Active Comparator)
  Interventions: Biological: AVX601
- C2 (Placebo Comparator)
  Interventions: Biological: Placebo
- T3 (Active Comparator)
  Interventions: Biological: AVX601
- C3 (Placebo Comparator)
  Interventions: Biological: AVX601
- T4 (Active Comparator)
  Interventions: Biological: AVX601
- C4 (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AVX601 — 3 doses of AVX601 at 1e7 IU given at T=0, 8, 24 weeks via the IM route
  Arms: T1
Biological: Placebo — 3 doses of placebo given at T=0, 8, 24 weeks via the IM route
  Arms: C1
Biological: AVX601 — 3 doses of AVX601 at 1e7 IU given at T=0, 8, 24 weeks via the SC route
  Arms: T2
Biological: Placebo — 3 doses of placebo given at T=0, 8, 24 weeks via the SC route
  Arms: C2
Biological: AVX601 — 3 doses of AVX601 at 1e8 IU given at T=0, 8, 24 weeks via the IM route
  Arms: T3
Biological: AVX601 — 3 doses of placebo given at T=0, 8, 24 weeks via the IM route
  Arms: C3
Biological: AVX601 — 3 doses of AVX601 at 1e8 IU given at T=0, 8, 24 weeks via the SC route
  Arms: T4
Biological: Placebo — 3 doses of placebo given at T=0, 8, 24 weeks via the SC route
  Arms: C4

SUMMARY:
AVX601, a bivalent alphavirus replicon vaccine expressing three CMV proteins (gB, pp65 and IE1) is a candidate vaccine against cytomegalovirus (CMV).

The objectives of this Phase 1 study are to test the safety of the vaccine and the immune response to the vaccine in healthy volunteers who have not previously been infected with CMV. Volunteers will be assigned by randomization to receive either the vaccine or an inactive substance (placebo) by injections in each arm on three occasions over 6 months. The study will last 12 months and will have a total of 12 visits.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled Phase 1 study of the safety and immunogenicity of AVX601 vaccine at two dosage levels and two routes of administration in healthy volunteers conducted at a single research center. A total of 40 participants will be enrolled into two groups of 20 participants each. Within each group, participants will be randomized to receive the active vaccine by IM injection (N = 8) or SC injection (N = 8) or to receive a placebo by IM injection (N = 2) or SC injection (N = 2). Each participant will receive a total of six injections of vaccine or placebo, two at each visit at Weeks 0, 8 and 24, administered by a study nurse in an outpatient setting, and will be followed for 12 months after the first immunization. Safety data will include local and systemic reactogenicity after each dose of vaccine, collected in a systematic format using a subject memory aid and a standard grading scale, specific safety laboratory parameters and general AEs. Immunogenicity data will be obtained by collecting blood at defined time points before and after immunization and separating serum (for measurement of antibodies to CMV by ELISA and neutralization assays and to the vaccine vector by a VRP neutralization assay) and peripheral blood mononuclear cells (PMBC) (for measurement of cellular immune responses to CMV peptides).

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 45 years of age, inclusive
2. Good general health without significant physical examination findings or clinically significant abnormal laboratory results
3. Available to participate for the entire study period of approximately 12 months
4. For women of childbearing potential, a negative urine pregnancy test at screening and before each immunization, and agreement to consistently use contraception from 28 days prior to enrollment until the last protocol visit, for sexual activity that could lead to pregnancy
5. Acceptable laboratory parameters:

   * negative CMV serology
   * hemoglobin ≥ 11.2 g/dL for women, ≥ 12.8 g/dL for men
   * white blood cell count 3,300 - 12,000 cells/mm3
   * platelet count 125,000 - 550,000/mm3
   * alanine aminotransferase (ALT) within normal range for study laboratory
   * serum creatinine within normal range for study laboratory
   * normal urine dipstick (negative glucose, negative hemoglobin, and negative or trace protein)
   * negative hepatitis B virus (HBV) and hepatitis C virus (HCV) blood tests
   * negative HIV blood test
6. Willingness to have blood stored for up to 10 years for use in additional assays to evaluate immune responses to CMV or the alphavirus vector if such assays become available
7. Willingness to participate in the study as evidenced by signed informed consent obtained before screening

Exclusion Criteria:

1. Venous access deemed inadequate for the phlebotomy demands of the study
2. Women who are breast feeding
3. In female subjects, a positive urine pregnancy test at screening or on the day of any vaccine injection
4. Receipt of any vaccine within 30 days prior to enrollment
5. Use of any investigational agent within 30 days prior to enrollment
6. Receipt of immunoglobulin or blood products within 60 days prior to enrollment
7. Use of cytotoxic medications within 6 months prior to enrollment
8. Use of systemic corticosteroids within 6 months prior to enrollment (except that participants who have completed a course of prednisone, at up to 20 mg per day for up to 7 days, at least 1 month prior to enrollment are eligible for enrollment)
9. History of serious adverse reactions to any vaccine, including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema or abdominal pain
10. History of immunodeficiency or autoimmune disease
11. History of diabetes mellitus
12. History of splenectomy
13. History of malignancy within the last 3 years (except that participants with a diagnosis of basal cell carcinoma of the skin are eligible for enrollment)
14. Psychiatric condition that may interfere with the ability to comply with the protocol requirements. Specifically excluded are persons with history of psychosis within the past 3 years or history of suicidal attempt or gesture within the past 3 years.
15. History of medical, occupational or family problems as a result of alcohol or illicit drug use during the past 12 months
16. Any condition which leads the investigator to believe that the participant cannot comply with the protocol requirements or that may place the participant at an unacceptable risk for participation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
evaluate safety of AVX601 based on teh frequency of Grade 2,3,or 4 systemic reactogenicity events | 1 year

SECONDARY OUTCOMES:
evaluate the immunogenicity of AVX601 in healthy volunteers after 3 doses of vaccine | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Olmsted, Ph.D., Principal Investigator — AlphaVax, Inc.
Locations (1):
- Cincinnati Center for Clinical Research, Cincinnati, Ohio, United States

REFERENCES:
- See also: AlphaVax Human Vaccines, Inc. — http://www.alphavax.com